CLINICAL TRIAL: NCT00126802
Title: The Role of Tomotherapy (Dynamic IMRT and Megavoltage CT Scanning) in Hypofractionated/Dose Escalated Conformal Radiation Treatment Using Magnetic Resonance Spectroscopy (MRS) Scans to Predict and Document the Pattern of Local Failure for High Risk Prostate Cancer
Brief Title: The Role of Tomotherapy in Hypofractionated/Dose Escalated Conformal Radiation Treatment for High Risk Prostate Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GU-06-0052/ethics 21781
Record Dates: First submitted 2005-08-03; First posted 2005-08-05 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: tomotherapy; MRSZ; high risk prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Tomotherapy — Standard 45 Gy in 25 fractions in 5 weeks

SUMMARY:
Helical tomotherapy is being used to treat the prostate gland, local rates of spread and regional lymph nodes whilst sparing gross structures. The radiation to the gross disease in the prostate is hypofractionated and dose escalated. Magnetic resonance spectroscopic imaging (MRSI) is incorporated into pre- and post-treatment evaluation.

ELIGIBILITY:
Inclusion Criteria:

* High risk localized prostate cancer

Exclusion Criteria:

* Low/intermediate risk, metastatic cancer
* Patient refusal

Max Age: 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-04; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Rectal Toxicity | 5 weeks
  Determine the acute and late rectal toxicity of high-dose short-course hypofractionated radiotherapy in five weeks in the treatment of high rish prostate cancer.

SECONDARY OUTCOMES:
prostate-specific antigen (PSA) and MRSI disease control | 3 years
  Determine the biochemical control (freedom from PSA failure) rate, overall and disease free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Pearcey, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada